CLINICAL TRIAL: NCT07392333
Title: A Prospective Cohort Study of Basivertebral Nerve Ablation Using the Stryker OptaBlate BVN System for the Treatment of Vertebrogenic Low Back Pain
Brief Title: Prospective Study of Basivertebral Nerve Ablation With the OptaBlate BVN System for Vertebrogenic Low Back Pain
Acronym: OptaBlate BVN
Status: Not yet recruiting | Type: Observational
Sponsor: Stryker Instruments (Industry)
Responsible Party: Sponsor
Other Study IDs: SISBVN12025US
Record Dates: First submitted 2026-01-26; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Verteborgenic Low Back Pain; Back Pain Lower Back
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- OptaBate BVN cohort
  Interventions: Device: Basivertebral nerve ablation

INTERVENTIONS:
Device: Basivertebral nerve ablation — The basivertebral nerve ablation is a minimally invasive, image-guided procedure in which radiofrequency energy is used to ablate the basivertebral nerve within the vertebral body, interrupting pain signals associated with vertebrogenic low back pain.

SUMMARY:
The goal of this observational study is to evaluate patient outcomes following treatment of vertebrogenic low back pain using the Stryker OptaBlate BVN System. Patients treated in accordance with the device IFU as part of routine clinical care and who consent to participate will be followed for 12 months after the procedure to assess treatment outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patient scheduled for treatment with the OptaBlate BVN System in accordance with the device IFU and willing to participate in the clinical investigation, undergo study procedure, engage in follow-up, able to read, write, speak, and understand English, and able to provide written informed consent.

Exclusion Criteria:

* The patient meets one or more contraindications as defined in the locally applicable IFU
* Spinal fracture or history of spinal trauma at index levels
* Previous lumbar fusion at any level
* Prior basivertebral nerve ablation at the target levels
* Vertebral cancer, spinal metastasis or Tumor-related vertebral fractures
* History of Osteoporotic vertebral fractures
* Spine interventions, including epidural steroid injections within 30 days
* BMI > 40 kg/m²
* Symptomatic spinal stenosis
* Radicular pain or leg pain greater than back pain
* Pregnancy or planning pregnancy during study period
* Enrollment in another interventional clinical trial
* Contraindication to MRI
* Life expectancy of less than 12 months

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic low back pain of at least 6 months' duration that has not responded to at least 6 months of conservative treatment and who demonstrate Type 1 or Type 2 Modic changes on MRI consistent with vertebrogenic pain.
Sampling Method: Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2026-03-31 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-11-30 (Estimated)

PRIMARY OUTCOMES:
Change in functional disability, assessed by the mean improvement in Oswestry Disability Index (ODI) score | 3 months post-procedure
Incidence and severity of adverse events related to the procedure and/or device. | 12 months post-procedure

SECONDARY OUTCOMES:
Change in ODI | 6 and 12 months post-procedure
Change in Visual Analogue Score (VAS) | 3, 6 and 12 months post-procedure
Rate of patients achieving clinical success at 3 months, defined as ODI improvement ≥10 points and VAS reduction ≥2 cm | 3 months post-procedure
Change in health-related quality of life (36-item Short Form Survey Instrument (SF-36)) | 3, 6, and 12 months post-procedure
Change in Pain Medication Dosage for Low Back Pain as Measured by Prescription Dosage Records | 3, 6 and 12 months post-procedure
Rate of additional procedures (lumbar transforaminal epidural steroid injections, lumbar interlaminar steroid injections, radiofrequency ablations etc.) | 12 months post-procedure
Imaging assessment - Magnetic Resonance Imaging (MRI) including Mean size of the lesion Rate of subjects with radiographic evidence of targeting success based on lesion location on MRI | 6 weeks post-procedure
Change in health-related quality of life (European Quality of Life 5 Dimensions 5 Level Version (EQ-5D-5L)) | 3, 6 and 12 months post-procedure
Assessment of global patient satisfaction | 3, 6 and 12 months post-procedure

CONTACTS AND LOCATIONS:
Locations (1):
- Cantor Spine Center, Fort Lauderdale, Florida, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared to protect patient confidentiality and because data sharing is not included in the informed consent or study protocol